CLINICAL TRIAL: NCT06742450
Title: Prospective Study of Constant Current Versus Constant Voltage Deep Brain Stimulation in Patients with Parkinson's Disease
Brief Title: Constant Current Versus Constant Voltage Subthalamic Nucleus Deep Brain Stimulation in Patients with Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Pins Medical Co., Ltd (Industry); Chinese PLA General Hospital (Other); Tianjin Huanhu Hospital (Other); Kunming Sanbo Brain Hospital (Unknown); Xijing Hospital (Other); The First People's Hospital of Changde City (Other); The General Hospital of Southern Theater Command (Other); THE FIRST AFFILIATED HOSPITAL OF SHIHEZI UNIVERSITY (Unknown); RenJi Hospital (Other); Changshu Hospital of Traditional Chinese Medicine (Other); Hainan General Hospital (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Second Affiliated Hospital of Bengbu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PX2024032
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Parkinson's Disease (PD)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Constant current (CC) subthalamic nucleus deep brain stimulation (Experimental)
  Interventions: Other: Constant current (CC) subthalamic nucleus deep brain stimulation
- Constant voltage (CV) subthalamic nucleus deep brain stimulation (Active Comparator)
  Interventions: Other: Constant voltage (CV) subthalamic nucleus deep brain stimulation

INTERVENTIONS:
Other: Constant current (CC) subthalamic nucleus deep brain stimulation — For subjects who have decided to undergo STN-DBS surgery and meet the inclusion criteria, the constant current (CC) mode is selected as the original electronic modality one week after surgery. Regardless of any changes in programming parameters over the following year, the constant current (CC) mode will be maintained.
  Arms: Constant current (CC) subthalamic nucleus deep brain stimulation
Other: Constant voltage (CV) subthalamic nucleus deep brain stimulation — For subjects who have decided to undergo STN-DBS surgery and meet the inclusion criteria, the constant voltage (CV) mode is selected as the original electronic modality one week after surgery. Regardless of any changes in programming parameters over the following year, the constant voltage (CV) mode will be maintained.
  Arms: Constant voltage (CV) subthalamic nucleus deep brain stimulation

SUMMARY:
To compare the efficacy, programming burden, power consumption, and physicians' and patients' satisfaction between current mode and voltage mode of deep brain stimulation in each period one year after surgery.

DETAILED DESCRIPTION:
This is a randomized, parallel controlled, multi-center study to compare the efficacy, programming burden, power consumption, and physicians' and patients' satisfaction between current mode and voltage mode of deep brain stimulation in each period one year after surgery. Participants will be followed for up to 12 months. Approximately 180 PD participants will be recruited from up to 14 sites. Participants will be randomized to current mode or voltage mode after DBS surgery and be comprehensively assessed at baseline and follow up according to the protocol developed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease
* Aged 18 to 75, no limited sex
* After bilateral STN-DBS, yet not powered on

Exclusion Criteria:

* Mental disorders or dementia
* Pregnant, lactating women or women who are unable to take effective measures to prevent pregnancy
* Serious health conditions, such as tumors, liver or kidney diseases, etc.
* Epilepsy or other seizure disorders
* Patients with severely deviated electrode placement
* Patients who were unable to voluntarily sign an informed consent form
* Patients who did not agree to cooperate with follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-01-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The change rate of MDS-UPDRS III | from baseline to 6 months after surgery
  MDS-UPDRS III is the motor examination section of the MDS-UPDRS (Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale), completed by the evaluator, providing an objective assessment of motor symptoms in patients with Parkinson's disease. MDS-UPDRS III ranges from 0-132. The change rate of MDS-UPDRS III in the Stim-On/Med-On state from baseline to 6 months after surgery will be collected. Positive indicates improvement.

SECONDARY OUTCOMES:
MDS-UPDRS I | from baseline to 6 months after surgery
  MDS-UPDRS I is the non-motor experiences of daily living section of the MDS-UPDRS (Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale). Subsection IA is evaluated by the researcher based on all relevant information provided by the patient or their caregiver regarding certain symptoms. Subsection IB is completed by the patient, with assistance from the caregiver if needed, but it must not be completed by the researcher. The change rate of MDS-UPDRS I from baseline to 6 months after surgery will be collected.
MDS-UPDRS II | from baseline to 6 months after surgery
  MDS-UPDRS II is the motor experiences of daily living section of the MDS-UPDRS (Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale) and is a self-reported questionnaire completed by the patient. The change rate of MDS-UPDRS II from baseline to 6 months after surgery will be collected.
MDS-UPDRS IV | from baseline to 6 months after surgery
  MDS-UPDRS IV is the motor complications section of the MDS-UPDRS (Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale). This section is rated by the evaluator, combining information provided by the patient with the evaluator's clinical observation and judgment to generate a comprehensive score. The change rate of MDS-UPDRS IV from baseline to 6 months after surgery will be collected.
Clinical Global Impression (CGI) | from baseline to 6 months after surgery
  The Clinical Global Impression (CGI) is a global assessment scale initially designed by the World Health Organization (WHO) for use in IPSS research to evaluate clinical efficacy. It provides an overall measure of treatment outcomes.
Physician satisfaction feedback | from baseline to 6 months after surgery
  The programming physician completes a custom-made questionnaire based on their subjective judgment.
Patient satisfaction feedback | from baseline to 6 months after surgery
  The patient completes a custom-made questionnaire based on their subjective judgment.
power consumption | from baseline to 6 months after surgery
  The total power consumption of the patient's IPG between visits is calculated. During follow-up, device logs are uploaded from the charging equipment to the database. The raw data is then retrieved from the database.
impecence | from baseline to 6 months after surgery
  Use the programming device to measure impedance on all contacts of the IPG.
Adverse effects | from baseline to 12 months after surgery
  Record any adverse events and serious adverse events during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes